CLINICAL TRIAL: NCT06565702
Title: Clinical Trial on the Accuracy of Blood Pressure Measurement by YE990 Medical Automatic Electronic Sphygmomanometer
Status: Not yet recruiting | Type: Observational
Sponsor: The First Affiliated Hospital of Anhui Medical University (Other)
Responsible Party: Principal Investigator, Hejun Liu, Chief Physician M.D., M.S., The First Affiliated Hospital of Anhui Medical University
Other Study IDs: YC20240201
Record Dates: First submitted 2024-07-15; First posted 2024-08-22 (Actual); Last update posted 2024-08-22 (Actual); Status verified 2024-08

CONDITIONS: Blood Pressure
Keywords: accuracy; systolic blood pressure; diastolic blood pressure; pulse rate; 12 years of age or older; automatic electronic sphygmomanometers

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Test medical equipment (blood pressure monitor): Name of device: Medical automatic electronic sphygmomanometer (Model: YE990) Registrant name: Jiangsu Yuyue Medical Equipment Co. Registration Certificate No.: Su Meizhi Quasi 20222071271 The minimum number of valid cases for the evaluation of the electronic sphygmomanometer with auscultation as a control, with sequential measurements in the same arm, was 85, of which 3 valid data sets were provided by each subject, for a total of 255 data sets.
- Control medical devices (reference sphygmomanometer): Name of device: Sphygmomanometer - stethoscope health care box (Model: A type) Registrant name: Jiangsu Yuyue Medical Equipment Co. Certificate of Registration No.: SuMeChiQi 20152070947 The minimum number of valid cases for the evaluation of the electronic sphygmomanometer with auscultation as a control, with sequential measurements in the same arm, was 85, of which 3 valid data sets were provided by each subject, for a total of 255 data sets.

SUMMARY:
This study was a single-center, open-ended, self-controlled clinical study . Same armsequential method was used to measure the blood pressure of the subjects，inclusion of ≥85 subjects aged 12 years or older who met the enrollment criteria.In accordance with the "Association for the Advancement of Medical Instrumentation/European Society of Hypertension/International Organization for Standardization (AAMI/ESH/ISO) Universal Standard (ISO 81060-2:2018/Amd 1:2020)",the purpose of this study was to compare the blood pressure and pulse rate measured by an electronic sphygmomanometer with those measured by a reference sphygmomanometer (an upper-arm noninvasive auscultatory sphygmomanometer) and by palpation of the radial artery, and then to evaluate the accuracy and safety of the measurement of systolic blood pressure, diastolic blood pressure, and pulse rate by a fully automated electronic sphygmomanometer for medical use (Model No. YE990), which is manufactured by Jiangsu Yuyue Medical Equipment Co.

DETAILED DESCRIPTION:
This study was a single-center, open-ended, self-controlled clinical study . Same armsequential method was used to measure the blood pressure of the subjects，inclusion of ≥85 subjects aged 12 years or older who met the enrollment criteria.In accordance with the "AAMI/ESH/ISO Universal Standard (ISO 81060-2:2018/Amd 1:2020)",the purpose of this study was to compare the blood pressure and pulse rate measured by an electronic sphygmomanometer with those measured by a reference sphygmomanometer (an upper-arm noninvasive auscultatory sphygmomanometer) and by palpation of the radial artery, and then to evaluate the accuracy and safety of the measurement of systolic blood pressure, diastolic blood pressure, and pulse rate by a fully automated electronic sphygmomanometer for medical use (Model No. YE990), which is manufactured by Jiangsu Yuyue Medical Equipment Co.

(One） criteria for admission Inclusion Criteria

Subjects should meet all of the following requirements for inclusion in the study:

1. Both sexes; at least 30% of the subjects are male and at least 30% of the subjects are female.
2. Subject's age > 12 years.
3. Arm circumference distribution:

   1. At least 20% of the subjects should have arm circumference within each quarter interval of the total arm circumference range;
   2. At least 10% of the subjects should have arm circumference within the upper one-eighth interval of the total arm circumference range;
   3. At least 10% of the subjects shall have an arm circumference within the lower one-eighth interval of the total arm circumference range.
4. Blood pressure distribution:

   1. At least 5% of subjects shall have a systolic blood pressure ≤100 mmHg (13.33 kPa);
   2. At least 5% of subjects shall have a systolic blood pressure ≥ 160 mmHg (21.33 kPa);
   3. At least 20% of subjects should have a systolic blood pressure ≥ 140 mmHg (18.66 kPa);
   4. Diastolic blood pressure should be ≤60 mmHg (8.0 kPa) in at least 5% of subjects;
   5. Diastolic blood pressure should be ≥100 mmHg (13.33 kPa) in at least 5% of subjects; (f) At least 20% of subjects should have a diastolic blood pressure ≥85 mmHg (11.33 kPa);
5. Subjects must be willing and able to comply with the study procedures by signing an informed consent form after being informed about the study.

consent form after understanding the contents of the study. (6) Good compliance and ability to complete the clinical trial. 2. Exclusion Criteria

Subjects who fulfill any of the following requirements cannot be included in the study:

1. Mental illness, impaired consciousness, or other conditions that prevent them from cooperating with the study;
2. Require hemodialysis;
3. Taking anticoagulant drugs for cardiovascular diseases;
4. Pregnant and lactating women;
5. Patients with cardiac arrhythmia;
6. Patients with peripheral arterial disease and diseases that may affect arterial compliance;
7. Other conditions that are considered by the physician to be unsuitable for enrollment.

（Two）Evaluation methods 2.1. Evaluation of effectiveness According to the standard requirements of "AAMI/ESH/ISO Universal Standard (ISO 81060-2:2018/Amd 1:2020)", the relationship between the mean value of the error and the standard deviation, the consistency between the measured and reference blood pressure values, and the relationship between the arm circumference and the measurement error should be evaluated.

1. Error mean and standard deviation Calculate the mean and standard deviation of the difference (i.e. error) between the measured and reference blood pressure values, and the result shall meet the requirements of ISO 81060-2:2018/Amd 1:2020 5.4.1.2.
2. Agreement between measured and reference blood pressure values (Bland-Altman analysis) For each measurement position, a scatter plot of the difference between the investigator and the device under test is obtained for each comparison of the investigator and the device under test, and the values of systolic and diastolic blood pressures shall be plotted separately.
3. Relationship between arm circumference and measurement error (Bland-Altman analysis) The relationship between upper arm circumference and measurement error is shown by plotting a scatter plot.
4. Relative pulse rate error Descriptive statistics of relative error in pulse rate.

2.2. Safety evaluation According to the "Code for Quality Management of Clinical Trials of Medical Devices" (2022) iii, medical devices should be collected and recorded when conducting clinical trials.

When conducting clinical trials of medical devices, the occurrence of adverse events and defects of the devices in the course of use by the subjects should be collected and recorded.

1. Incidence of adverse events;
2. Incidence of device defects.

2.3. Evaluation of product performance Clinical use performance evaluation is mainly for product stability evaluation, the specific evaluation criteria are as follows, the following items if evaluation

If the evaluation of the following items is "yes", it is necessary to specifically describe the cause of the failure:

Evaluation item 1: electronic sphygmomanometer power on and off Yes: Cannot be turned on and/or off normally; No: can be turned on and off normally. Evaluation Item II: Whether the device automatically shuts off during the checking process Yes: Automatic shutdown during the inspection; No: There is no automatic shutdown during the inspection. Evaluation item 3: Whether there is any abnormal interruption due to the machine during the inspection process.

Yes: Abnormal interruptions occurred during the inspection process due to the machine; No: No abnormal interruptions occurred during the inspection. Evaluation item 4: Whether inflation and exhaust failures occurred during the inspection process Yes: Inflation and/or exhaust failure occurred during the inspection; No: No inflation and exhaust failure occurred during the inspection. Evaluation item 5: Whether air leakage occurred during the inspection process Yes: Air leakage occurred; No: no air leakage occurred.

（Three）Test medical device and control medical device

1. Test medical equipment (blood pressure monitor) Name of device: Medical automatic electronic sphygmomanometer (Model: YE990) Registrant name: Jiangsu Yuyue Medical Equipment Co. Registration Certificate No.: Su Meizhi Quasi 20222071271
2. Control medical devices (reference sphygmomanometer) Name of device: Sphygmomanometer - stethoscope health care box (Model: A type) Registrant name: Jiangsu Yuyue Medical Equipment Co. Certificate of Registration No.: SuMeChiQi 20152070947

（Four）statistical analysis

1. General principles Descriptive statistical analysis: qualitative indicators are described by frequency tables and percentages; quantitative indicators are described by mean, standard deviation, minimum, median, maximum, upper quartile (Q1) and lower quartile (Q3).

2. Content of statistical analysis

1. The number of subjects enrolled, dislodged, and completed cases, and a list of reasons why subjects withdrew from the study.
2. Demographic and vital sign data of the subjects Quantitative data were analyzed by describing their number of cases, mean, standard deviation, minimum, median, maximum, and upper quartile.

   maximum, upper quartile (Q1), and lower quartile (Q3); qualitative data were analyzed by describing the number of cases and their proportion of the total number of subjects.

   The qualitative data were analyzed by describing the number of cases and their percentages.
3. Validity analysis Error mean and standard deviation According to ISO 81060-2:2018/Amd 1:2020 5.4.1.2, the error mean and standard deviation deviation should meet the following evaluation criteria: Criterion 1: Calculate the mean and standard deviation of the errors of the 255 groups of measured and reference blood pressure values for 85 subjects.

Criterion 1: Calculate the mean and standard deviation of the errors of 255 sets of measured and reference blood pressure values of 85 subjects, and compare the systolic and diastolic blood pressures separately, with the mean value of the error not exceeding ±5 mmHg and the standard deviation not exceeding 8 mmHg.

Criterion 2: Comparison of the mean of the three sets of errors for each subject, comparing systolic and diastolic blood pressures separately.

Agreement between measured and reference blood pressure values (Bland-Altman analysis) According to ISO 81060-2:2018/Amd 1:2020, a scatter plot of the difference between the reference device and the device under test should be plotted for each occasion, and the difference between systolic and diastolic blood pressure should be plotted separately. x-axis indicates the mean value of the 2 methods of measurement for each subject, and y-axis indicates the difference between the 2 methods of measurement for each subject.

Relationship between arm circumference and measurement error (Bland-Altman analysis) Plot the results of all subjects by arm circumference according to ISO 81060-2:2018/Amd 1:2020 5.1.4 d. The x-axis shows the actual arm circumference of the subject and the y-axis shows the difference between the measured blood pressure value and the reference blood pressure value.

Pulse Rate Error The relative error of the pulse rate measurement is counted.

ELIGIBILITY:
Inclusion Criteria:

Subjects should meet all of the following requirements for inclusion in the study:

1. Both sexes; at least 30% of the subjects are male and at least 30% of the subjects are female.
2. Subject's age > 12 years.
3. Arm circumference distribution:

   1. At least 20% of the subjects should have arm circumference within each quarter interval of the total arm circumference range;
   2. At least 10% of the subjects should have arm circumference within the upper one-eighth interval of the total arm circumference range;
   3. At least 10% of the subjects shall have an arm circumference within the lower one-eighth interval of the total arm circumference range.
4. Blood pressure distribution:

   1. At least 5% of subjects shall have a systolic blood pressure ≤100 mmHg (13.33 kPa);
   2. At least 5% of subjects shall have a systolic blood pressure ≥ 160 mmHg (21.33 kPa);
   3. At least 20% of subjects should have a systolic blood pressure ≥ 140 mmHg (18.66 kPa);
   4. Diastolic blood pressure should be ≤60 mmHg (8.0 kPa) in at least 5% of subjects;
   5. Diastolic blood pressure should be ≥100 mmHg (13.33 kPa) in at least 5% of subjects; (f) At least 20% of subjects should have a diastolic blood pressure ≥85 mmHg (11.33 kPa);
5. Subjects must be willing and able to comply with the study procedures by signing an informed consent form after being informed about the study.

   consent form after understanding the contents of the study.
6. Good compliance and ability to complete the clinical trial.

Exclusion Criteria:

Subjects who fulfill any of the following requirements cannot be included in the study:

(1) Mental illness, impaired consciousness, or other conditions that prevent them from cooperating with the study; (2) Require hemodialysis; (3) Taking anticoagulant drugs for cardiovascular diseases; (4) Pregnant and lactating women; (5) Patients with cardiac arrhythmia; (6) Patients with peripheral arterial disease and diseases that may affect arterial compliance; (7) Other conditions that are considered by the physician to be unsuitable for enrollment.

-

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Healthy people over 12 years of age who meet the criteria for admission to the platoon
Sampling Method: Probability Sample
Enrollment: 85 (Estimated)
Dates: Start 2024-08-20 (Estimated); Primary Completion 2025-08-20 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
To evaluate the accuracy of the arm-type electronic blood pressure monitor (Model: YE660D) in measuring systolic blood pressure, diastolic blood pressure and pulse rate in adults aged 12 years and above. | August 20, 2024 - December 30, 2025
  Evaluate the relationship between the mean and standard deviation of error, the agreement between the measured and reference blood pressure values, and the relationship between arm circumference and measurement error.Reference standard: 255 sets of data from 85 subjects were calculated and compared separately for systolic and diastolic blood pressure, with a mean deviation of not more than ±5 mmHg and a standard deviation of not more than 8 mmHg.

SECONDARY OUTCOMES:
Collect and document the occurrence of adverse events and device defects in subjects during use | August 20, 2024 - December 30, 2025
  1. Incidence of adverse events;
  2. Incidence of device defects.

OTHER OUTCOMES:
Clinical use performance evaluation is mainly product stability evaluation | August 20, 2024 - December 30, 2025
  Evaluation Item 1: Electronic Sphygmomanometer Turning On and Off Evaluation item 2: Whether the device was turned off automatically during the checking process Evaluation item 3: Whether there is any abnormal interruption due to the machine during the inspection process.
  Evaluation item 4: Whether inflation and exhaust failure occurs during the inspection process Evaluation item 5: Whether air leakage occurred during the inspection process

CONTACTS AND LOCATIONS:
Overall Officials: Hejun Liu, Principal Investigator — The First Affiliated Hospital of Anhui Medical University
Locations (1):
- The First Affiliated Hospital of Anhui Medical University Hospital, Hefei, Anhui, China

REFERENCES:
- [Derived] Xu D, Tang H, Wang C, Cheng H, Wu W, Lu Q, Liu H. Validation of the YuWell YE990 medical automatic electronic blood pressure monitor according to the Association for the Advancement of Medical Instrumentation/European Society of Hypertension/International Organization for Standardization Universal Standard (ISO 81060-2:2018/Amd.1:2020). Blood Press Monit. 2025 Aug 1;30(4):191-195. doi: 10.1097/MBP.0000000000000755. Epub 2025 May 6. PMID 40327332

DOCUMENTS (1):
  • Informed Consent Form (2024-04-15): https://cdn.clinicaltrials.gov/large-docs/02/NCT06565702/ICF_000.pdf